CLINICAL TRIAL: NCT06506630
Title: Effects of Coenzyme Q10 Supplement on Cardiovascular Risk Factors in Subjects at High Risk of Metabolic Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tian Zezhong (Other)
Responsible Party: Sponsor-Investigator, Tian Zezhong, Research Fellow, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20240703
Record Dates: First submitted 2024-07-03; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Metabolic Syndrome; Cardiovascular Diseases
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CoQ10 1R (Placebo Comparator): take orally 600 mg placebo per day
  Interventions: Dietary Supplement: placebo
- CoQ10 2R (Experimental): take orally 600 mg drug per day (contains 100mg coenzyme Q10)
  Interventions: Dietary Supplement: coenzyme Q10
- CoQ10 3R (Experimental): take orally 600 mg drug per day (contains 200mg coenzyme Q10)
  Interventions: Dietary Supplement: coenzyme Q10

INTERVENTIONS:
Dietary Supplement: coenzyme Q10 — 300 mg capsule twice a day
  Arms: CoQ10 2R; CoQ10 3R
Dietary Supplement: placebo — 300 mg capsule twice a day
  Arms: CoQ10 1R

SUMMARY:
This study aims to evaluate the ameliorating effect of coenzyme Q10 supplementation on cardiovascular risk factors in high risk population for metabolic syndrome, including blood lipid metabolism, insulin resistance, blood pressure regulation, platelet function, endothelial function, cardiorespiratory fitness and muscle function.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome or high-risk groups with metabolic syndrome are defined as subjects with metabolic syndrome according to the International Diabetes Federation (IDF) Chinese Adult Criteria, and high-risk groups are defined as those who meet at least two MetS risk factors. The specific criteria are as follows:

  1. Aged 30-90 years old;
  2. Two or more of following are acceptable:

  <!-- -->

  1. Abdominal obesity (central obesity): waist circumference >=90 cm for men and >=80cm for women;
  2. Hyperglycemia: fasting blood glucose ≥ 5.6mmol/L or taking hypoglycemic drugs;
  3. Hypertension: systolic blood pressure >=130mmHg and (or) diastolic blood pressure >=85mmHg or taking blood pressure medications;
  4. Fasting TG>=1.70mmol/L or taking antihyperlipidemic drug;
  5. Fasting HDL-C<1.04 mmol/L for men, <1.29 mmol/L for women or taking antihyperlipidemic drug; 3) Sign informed consent and insist on participating in the research.

Exclusion Criteria:

* 1) Take drugs/dietary supplements, such as aspirin, fish oil and etc., that affect platelet function in recently six months; 2) blood system disease or infection; 3) Blood pressure >=160/100mmHg; 4) Low platelet count (whole blood platelet<100 x 10^9/mL); 5) Abnormal hemoglobin (male <120g/L, female <110g/L); 6) Low hematocrit (male <40%, female <37%); 7) Prothrombin time (PT) is outside the normal reference range; 8) Pregnant women or nursing mothers; 9) Abnormal menstrual cycle, taking birth control pills or hormone replacement therapy; 10) Gastric ulcer, liver or kidney dysfunction.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
platelet aggregation | baseline and week 24
  Fresh PRP prepared from subjects was stimulated by ADP at baseline and at 24 weeks. Platelet aggregation was evaluated on a Chronolog aggregometer (Chrono-Log Corp., PA, USA) in PRP (3.0 × 10^8 platelets/mL) at 37 °C, and the change in light transmission was monitored and recorded for at least 5 minutes.
platelet acativation | baseline and week 24
  freshly isolated PRP was separately incubated with different fluorescent-labeled antibodies activated GPⅡbⅢa (FITC-conjugated mouse anti-human PAC-1) or P-selectin (FITC-conjugated mouse anti-human CD62P) at room temperature for 30 min. Platelets were initiated by adding 100 µmol/L adenosine diphosphate (ADP) at room temperature, followed by fixation with 1% paraformaldehyde (pH = 7.2) before analysis. All samples were analyzed via a calibrated CytoFLEX flow cytometer.
Platelet granule release | baseline and week 24
  using Elisa kits to detect PF4, β-TG, RANTES, TGF-β1 and soluble P-selectin (sP-selectin) levels
cardiorespiratory fitness | baseline and week 24
  using a comprehensive set of tests including spirometry for lung function, Incremental load test for exercise capacity, and a maximal oxygen uptake test (VO2 max) for aerobic fitness. Spirometry will quantify lung function by measuring forced vital capacity (FVC) and forced expiratory volume in one second (FEV1).
Change from Baseline in Muscle Mass to Week 24 | baseline and week 24
  Muscle mass was measured by bioelectrical impedance analysis with the use of a body composition analyzer. Change = (Week 24 Muscle Mass - Baseline Muscle Mass).
Change from Baseline in Handgrip Strength to Week 24 | baseline and week 24
  Handgrip strength was measured by a hand dynamometer following a standardized procedure. Change = (Week 24 Handgrip Strength - Baseline Handgrip Strength).
Change from Baseline in Usual Gait Speed to Week 24 | baseline and week 24
  Usual gait speed was measured by the 6-metre walk test following a standardized procedure. Change = (Week 24 Usual Gait Speed - Baseline Usual Gait Speed).

SECONDARY OUTCOMES:
Blood pressure | baseline and week 24
  blood pressure will be assessed using a validated and calibrated sphygmomanometer. Blood pressure will be measured in millimeters of mercury (mmHg), with systolic and diastolic pressures recorded separately. Participants will be asked to rest for at least 5 minutes in a quiet environment before the measurement to ensure accuracy. The average of three consecutive readings, taken at 1-minute intervals, will be used to determine the participant's blood pressure.
Fasting blood sugar | baseline and week 24
  Fasting blood glucose will be measured in milligrams per deciliter (mg/dL) using the standard hexokinase method. Participants are required to fast for at least 8 hours before blood sampling, with the exception of water. The test will be carried out in a laboratory setting using a calibrated automatic biochemical analyzer.
Blood lipids profile | baseline and week 24
  including the assessment of six key components: total cholesterol (TC), triglycerides (TG), low-density lipoprotein cholesterol (LDL-C), high-density lipoprotein cholesterol (HDL-C), apolipoprotein A-I (Apo A-I) and B (Apo B). These measurements will be conducted using standard enzymatic assays in a clinical laboratory setting. Blood samples will be collected after an overnight fast of at least 8 to 12 hours. The results will be reported in milligrams per deciliter (mg/dL) for TC, TG, LDL-C, and HDL-CApo A-I and Apo B will be reported in grams per liter (g/L).

CONTACTS AND LOCATIONS:
Locations (1):
- School of Public Health (Shenzhen), Sun Yat-sen University, Shenzhen, China

IPD SHARING:
Plan to Share IPD: No